CLINICAL TRIAL: NCT00257842
Title: Randomized Controlled Trial of Biofeedback Therapy for Dyssynergic Defecation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, pi, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DK057100-05 (NIH)
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Dyssynergia
MeSH Terms: conditions — Ataxia | interventions — Biofeedback, Psychology

INTERVENTIONS:
Procedure: Standard treatment, sham feedback and biofeedback therapy

SUMMARY:
Constipation is a common disorder and current treatments are unsatisfactory. Biofeedback may help patients with constipation and dyssynergic defecation, but its efficacy is unproven and whether this is due to behavioral modification or excessive attention is unknown. Methods: In a prospective randomized trial, the investigators investigated the efficacy of Biofeedback (manometric- assisted anal relaxation, muscle coordination and simulated defecation training), with either sham feedback therapy (Sham) or standard therapy (diet, exercise, laxatives; Standard) in 77 subjects (69 women) with dyssynergic defecation. Primary outcome measures included presence of dyssynergia, balloon expulsion time, number of complete spontaneous bowel movements (CSBM), and global bowel satisfaction. Data analyzed per protocol.

ELIGIBILITY:
Inclusion Criteria:Patients were included if they fulfilled Rome II criteria for functional constipation, and during attempted defecation demonstrated a dyssynergic pattern of defecation, and either had prolonged difficulty with expelling a simulated stool (> 1 minute) or prolonged delay (> 20% marker retention) in colonic transit.

Exclusion Criteria: They were required to have no evidence of structural or metabolic diseases that could cause constipation, as assessed by colonoscopy/barium enema and routine hematological, biochemical and thyroid function tests. Patients taking drugs known to be constipating, for example opioids were either excluded or were asked to discontinue the drug prior to enrollment. Other exclusion criteria included: severe cardiac or renal disease, previous gastrointestinal, spinal or pelvic surgery except cholecystectomy, hysterectomy or appendectomy, neurologic diseases such as multiple sclerosis, stroke or spinal injury, impaired cognizance (mini-mental score < 15), legal blindness, pregnancy, rectal prolapse, anal fissure, and alternating constipation and diarrhea.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Satish SC Rao, MD, PhD., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States